CLINICAL TRIAL: NCT06191965
Title: Double Blind, Randomized, Placebo-Controlled Study of MitoQ as Adjunctive Treatment for Patients With Early-phase Schizophrenia-spectrum Disorder and Mitochondrial Dysfunction
Brief Title: MitoQ for Early-phase Schizophrenia-spectrum Disorder and Mitochondrial Dysfunction
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Yale University (Other); University of Lausanne (Other)
Responsible Party: Principal Investigator, Dost Ongur, Professor of Psychiatry/Psychotic Disorders Division Chief, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P000970
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia and Related Disorders; Mitochondrial Alteration; Cognitive Impairment
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction | interventions — mitoquinone; Sugars

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial of MitoQ vs. placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The person in charge of the randomization will manage a database with codes matched to the assigned treatment of each patient after the initial screening visit. Trial participants, clinicians, outcome assessors, and researchers involved in the assessments and analyses of collected data will remain blind concerning the MitoQ or placebo randomization. Unblinding is permissible at a clinician's request, for safety reasons, when the health condition of the participant may be or may have been affected by the administration of MitoQ or placebo. In such cases, study staff will find out from the person in charge of randomization which treatment the patient is receiving (MitoQ or placebo) and immediately communicate that information to the patient's clinician. After a participant's allocated intervention has been revealed, however, the subject will be excluded from the trial. The data collected to that point will be included in analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MitoQ (Experimental): 20 mg 2 capsules once daily for 12 weeks (total daily dose 40 mg)
  Interventions: Drug: MitoQ
- Placebo (Placebo Comparator): 2 capsules (identical in appearance to MitoQ capsules) once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MitoQ — MitoQ is a synthetic analogue of coenzyme Q10. It is produced by the company Antipodean Pharmaceuticals and is formulated as a stable yellow powder suitable for oral formulation, prepared as capsules of white color. It is a commercial dietary supplement sold over the counter as an antioxidant, to be taken orally once or twice a day. It has subsequently been tested for various clinical conditions in humans.
  1. Molecular formula: C38H47O7PS (C37H44O4P.CH3O3S)
  2. CAS number: 444890-41-9 (phosphonium cation)
  3. Molecular weight: 678.81
  4. MitoQ capsules: The standard commercial posology is a 20 mg daily dose. All formulations are produced following Good Manufacturing Practice (GMP) standards (https://www.who.int/medicines/areas/quality_safety/quality_assurance/TRS986annex2.pdf?ua=1).
  5. MitoQ will be administered in oral capsules provided by the manufacturer Antipodean Pharma, to be taken once daily, one hour before breakfast. The daily dose will be 2 pills, i.e., 40 mg MitoQ.
  Other Names: mitoquinol mesylate; Chemical name: [10-(4,5-dimethoxy-2-methyl-3,6-dioxo-1,4-cyclohexadien-1-yl) decyl] triphenyl phosphonium mesylate
  Arms: MitoQ
Drug: Placebo — Placebo pills in identical appearance to the MitoQ capsules will be produced and provided by Antipodean Pharma and given to the patients in the control arm two per day to be taken one hour before breakfast. The composition of the placebo is tapioca starch, microcrystalline cellulose, hypromellose, silica-colloidal anhydrous, purified water, carrageenan, and pectin.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The goal of this double-blind, placebo-controlled randomized clinical trial is to test the effect of 12 weeks of orally administered MitoQ (mitoquinol mesylate) supplementation on cognition in 50 people with early phase schizophrenia-spectrum disorders (E-SSD) who have mitochondrial dysfunction (called high risk, or HR). Cognitive impairments in SSD can cause significant disability. Yet, there are no effective treatments for cognitive impairments in SSD. It has been shown that alterations in a certain type of brain cell (parvalbumin interneurons, or PVI) underlie cognitive deficits in SSD. These PVI, which fire at a fast rate, utilize high amounts of energy from the mitochondria and are highly vulnerable to oxidative stress. MitoQ is an antioxidant. Research has shown that, in mice, MitoQ can reduce oxidative stress in the mitochondria. The main question that this clinical trial aims to answer is:

• Does MitoQ supplementation, compared to placebo, improve cognition in HR patients?

Secondary questions that this clinical trial aims to answer are the following: Does MitoQ supplementation, compared to placebo:

* Improve positive and negative symptoms of SSD in HR patients?
* Improve functioning in HR patients?
* Improve/normalize blood markers of mitochondrial dysfunction in HR patients?

The investigators will enroll 100 individuals with E-SSD. These enrolled participants will participate in an initial screening visit to determine if they qualify for the actual clinical trial. At the screening visit, the investigators will ask about psychiatric history to determine diagnosis; ask about medical history; do a physical exam; collect blood and urine samples; do a pregnancy test; and ask participants to bring in their current medications in their original packaging so it is known what they are taking.

After the screening visit, the investigators will invite 50 HR patients (identified with a blood test) to continue with the clinical trial. Participants who qualify for the clinical trial will be asked to:

* Take a supplement (MitoQ or placebo) once per day for 12 weeks in addition to their usual medications.
* Come in for a study visit every 4 weeks over the 16-week study period. At these study visits, the investigators will do a physical exam; ask about symptoms and side effects; take blood and urine samples; and ask questions about general health and well-being, quality of life, mental health, emotional health, and mood. At visits 1 (baseline) and 4 (12 weeks), participants will also take a cognitive assessment.

DETAILED DESCRIPTION:
The planned clinical trial aims to test the effect of an oral administration of MitoQ on neurocognition, psychiatric symptoms, functioning, and exosomal levels of the mechanism-based biomarkers miR-137 and COX6A2 in HR individuals in the early phase of schizophrenia-spectrum disorders (E-SSD).

The investigators propose to implement a randomized, double-blind, placebo-controlled stratified clinical trial with MitoQ as an adjunctive treatment for 12 weeks in a sample of n=25 patients with early-stage psychosis. The primary outcome will be a change in global cognition as defined by the MATRICS Consensus Cognitive Battery (MCCB). Specifically, the hypothesis is that MitoQ will lead to an increase in the MCCB cognitive composite score in the subgroup of early psychosis patients displaying peripheral markers of mitochondrial dysfunction.

To test whether the oral administration of MitoQ will improve neurocognition in the HR subgroup, the investigators will conduct a double-blind, randomized, placebo-controlled trial at two sites (McLean Hospital and Yale School of Medicine). The overall goal of the study is to assess 100 patients (50 per site) with early phase psychotic disorders for HR status (with a blood test) and randomize 50 HR patients (25 per site). This 50% proportion is based on the fact that, in the Early psychosis Lausanne Cohort, the HR patients constitute half of the entire cohort 1.

The two sites will conduct research procedures in parallel, following the same protocol, but undergo independent processes of human subjects review and oversight by each site's local institutional review board. Thus, at McLean (for which the Mass General Brigham IRB will serve as the IRB of record), the investigators plan to assess 50 early psychosis patients for HR status and randomize 25 HR patients to MitoQ vs. placebo. An equivalent number of participants will be enrolled and randomized at Yale (for which the Yale IRB will serve as the IRB of record). With 20% attrition, it is expected that there will be 20 completers per site at the end of the study.

Patients will be asked to take part in a clinical trial consisting of a randomization to either MitoQ or placebo for 12-weeks and a follow up visit 4 weeks after the end of the last intervention.

Patients who are in the first 5 years of treatment for a SCZ-spectrum disorder will be eligible 30. All eligible patients with an early phase psychotic disorder will be recruited for this study. Patients who enroll in the study will undergo a blood test during the screening visit to determine if their plasma mIR137 and COX6A2 levels are consistent with high risk (HR) or low risk (LR) status. Once this categorization has been made, only HR patients will be invited to proceed with the study. HR patients who wish to continue will be assigned randomly to either the MitoQ or the placebo arm.

Primary outcome:

- Our primary outcome is change in cognitive function, as measured by change in the composite MCCB score from baseline to 12 weeks.

Secondary outcomes:

* The investigators will also measure each specific neurocognitive domain within the MCCB because each domain includes differential information. For example, attention/vigilance appears to best differentiate HR from LR patients.
* The investigators will also include change in clinical outcomes and blood biomarkers as described in the sections below:

  1. Global Assessment of Functioning (GAF) and the Social and Occupational Functioning Assessment Scale (SOFAS)
  2. Positive and negative symptoms (Positive and Negative Syndrome Scale- PANSS)
  3. Blood biomarkers: Improvement/normalization of the exosomal levels of miR-137 and COX6A2 to demonstrate target engagement.
  4. Clinical global impression (CGI) score: Change in global illness severity, measured with the Clinical Global Impressions-Severity (CGI-S).

Safety Outcomes:

All adverse effects, vital signs, ED visits and hospitalizations, and the Generic assessment of side effects scale (GASE-D) score will be recorded at every visit. There will also be an EKG obtained at the screening visit, at the start of treatment (week 0), and at week 12.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 35 years old
* Patients who have been diagnosed with one of the following schizophrenia-spectrum disorders: schizophreniform disorder, schizophrenia, schizoaffective disorder, unspecified psychosis.
* Less than five years in treatment for psychosis (note that the duration of psychosis may be longer than 5 years, but this is more difficult to ascertain and therefore less reliable as an inclusion criterion).
* PANSS score < 75
* Ability to provide informed consent.

Exclusion Criteria:

* Meeting DSM-5 criteria for any substance use disorder diagnosis in the past 6 months will be exclusionary EXCEPT tobacco and mild/moderate cannabis use disorder, which will be included
* Any acute medical condition requiring actively changing treatment (e.g., autoimmune disorders, acute infections, HIV/AIDS, cancer, renal failure, hepatic dysfunction, cardiovascular disease, or abnormal thyroid findings). Individuals with chronic medical conditions that are stable will not be excluded (e.g., person with hypothyroidism who is taking thyroid hormone replacement and has TSH levels within the normal range; person with well-managed diabetes; etc.)
* Epilepsy or another seizure disorder
* Intellectual disability (e.g., history of IQ < 70).
* Under legal guardianship
* Not English speaking. The questionnaires, instruments, cognitive assessments used in this research study have not been translated, validated, or studied extensively in non-English-speaking individuals. For this reason, we will not enroll individuals who do not speak English to maintain validity in the study.
* MitoQ allergy
* Treatment with antioxidants: omega3 (fish oil), Vitamin E, Vitamin C, multivitamins, NAC (N-acetyl cysteine) within the last 14 days. If the treatment is taken without prescription, we will ask the patient to stop using it for at least 14 days to become eligible for the present study.
* Children and adolescents, pregnant women, women who have the intention to become pregnant during the course of the study, and breastfeeding women are excluded from the study. This is because no MitoQ pharmacokinetic data are available in pediatric populations, pregnancy or breastfeeding.
* Lack of safe contraception, defined as: female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases. Female participants who are surgically sterilized/hysterectomized or post-menopausal for longer than 2 years are not considered as being of childbearing potential.
* Enrollment of study staff, their family members, and other dependent persons

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the MATRICS Consensus Cognitive Battery (MCCB) composite score at week 12 | Baseline and week 12
  The MCCB evaluates cognitive functioning in schizophrenia and related disorders. It includes ten tests that measure seven cognitive domains including speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The MCCB composite score has been shown to be highly correlated with general level of intellectual ability.

SECONDARY OUTCOMES:
Change from baseline in the MATRICS Consensus Cognitive Battery (MCCB) attention/vigilance score at week 12 | Baseline and week 12
  The MCCB evaluates cognitive functioning in schizophrenia and related disorders. It includes ten tests that measure seven cognitive domains including speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. Research has suggested that the attention/vigilance domain best differentiates HR from low risk (LR) patients.
Change from baseline in the MATRICS Consensus Cognitive Battery (MCCB) speed of processing score at week 12 | Baseline and week 12
  The MCCB evaluates cognitive functioning in schizophrenia and related disorders. It includes ten tests that measure seven cognitive domains including speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition.
Change from baseline in the MATRICS Consensus Cognitive Battery (MCCB) working memory score at week 12 | Baseline and week 12
  The MCCB evaluates cognitive functioning in schizophrenia and related disorders. It includes ten tests that measure seven cognitive domains including speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition.
Change from baseline in the MATRICS Consensus Cognitive Battery (MCCB) verbal learning score at week 12 | Baseline and week 12
  The MCCB evaluates cognitive functioning in schizophrenia and related disorders. It includes ten tests that measure seven cognitive domains including speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition.
Change from baseline in the MATRICS Consensus Cognitive Battery (MCCB) visual learning score at week 12 | Baseline and week 12
  The MCCB evaluates cognitive functioning in schizophrenia and related disorders. It includes ten tests that measure seven cognitive domains including speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition.
Change from baseline in the MATRICS Consensus Cognitive Battery (MCCB) reasoning and problem solving score at week 12 | Baseline and week 12
  The MCCB evaluates cognitive functioning in schizophrenia and related disorders. It includes ten tests that measure seven cognitive domains including speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition.
Change from baseline in the MATRICS Consensus Cognitive Battery (MCCB) social cognition score at week 12 | Baseline and week 12
  The MCCB evaluates cognitive functioning in schizophrenia and related disorders. It includes ten tests that measure seven cognitive domains including speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition.
Change from baseline in the Positive and Negative Syndrome Scale (PANSS) total score at week 12 | Baseline and week 12
  The PANSS is a 30-item clinician-administered rating scale that evaluates the severity of positive, negative, and general psychopathology symptoms in schizophrenia and related psychotic disorders. Each of the 30 items is rated from 1 to 7, ranging from absent to extreme. The total PANSS score, which is the sum of the three subscales ranges from 30 to 210 (7-49 for the positive scale, 7-49 for the negative scale, and 16-112 for the general psychopathology scale).
Change from baseline in the Social and Occupational Functioning Assessment Scale (SOFAS) score at week 12 | Baseline and week 12
  The SOFAS is a global rating of current functioning ranging from 0 to 100, with lower scores representing lower functioning. The SOFAS differs from the similar Global Assessment of Functioning (GAF) scale by focusing on social and occupational functioning independent of the overall severity of the individual's psychological symptoms. The SOFAS also differs from the GAF scale in assessing impairments in functioning due to physical limitations, as well as those due to mental impairments.
Change from baseline in the Global Assessment of Functioning (GAF) score at week 12 | Baseline and week 12
  The GAF score is used to rate how serious a mental illness may be. It measures how much a person's symptoms affect their day-to-day life on a scale of 0 to 100, with lower scores representing lower functioning.
Change from baseline in the Clinical Global Impressions Severity (CGI-S) scale score at week 12 | Baseline and week 12
  The CGI-Severity (CGI-S) scale asks the clinician one question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. This rating is based upon observed and reported symptoms, behavior, and function in the past seven days.
Change from baseline in the level of miR-137 at week 12 | Baseline and week 12
  miR-137 (or microRNA-137) is a short exosomal (non-coding) RNA molecule that functions to regulate the expression levels of other genes. mIR-137 is a marker of mitochondrial dysfunction in early psychosis (with higher levels associated with greater mitochondrial dysfunction). Changes in mIR-137 in combination with changes in COX6A2 will help us determine the success of target engagement.
Change from baseline in the level of COX6A2 at week 12 | Baseline and week 12
  The protein COX6A2 is a subunit of cytochrome c oxidase complex IV specific to parvalbumin interneurons, which are known to be altered in schizophrenia. COX6A2 is a marker of mitochondrial dysfunction in early psychosis (with lower levels associated with greater mitochondrial dysfunction). Changes in COX6A2 in combination with changes in mIR-137 will help us determine the success of target engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Dost Ongur, MD, PhD, Principal Investigator — Mclean Hospital
Locations (3):
- United States (2):
  - Yale School of Medicine, New Haven, Connecticut
  - McLean Hospital, Belmont, Massachusetts
- University of Lausanne, Lausanne, Switzerland

REFERENCES:
- [Background] Khadimallah I, Jenni R, Cabungcal JH, Cleusix M, Fournier M, Beard E, Klauser P, Knebel JF, Murray MM, Retsa C, Siciliano M, Spencer KM, Steullet P, Cuenod M, Conus P, Do KQ. Mitochondrial, exosomal miR137-COX6A2 and gamma synchrony as biomarkers of parvalbumin interneurons, psychopathology, and neurocognition in schizophrenia. Mol Psychiatry. 2022 Feb;27(2):1192-1204. doi: 10.1038/s41380-021-01313-9. Epub 2021 Oct 22. PMID 34686767